CLINICAL TRIAL: NCT03567161
Title: Ultrasonic Surgical Aspirator to Treat Deep Infrabony Defects: A New Flapless Minimally Invasive Approach
Brief Title: Ultrasonic Surgical Aspirator to Treat Deep Infrabony Defects
Acronym: CUSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giovanni Lodi, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CUSA
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cavitron ultrasonic surgical aspirator (Experimental): Patients.with periodontitis.
  Inclusion criteria:
  1. Having received a diagnosis of chronic periodontitis (Armitage 1999)
  2. Being treated by full mouth debridement, and supportive periodontal treatment (SPT) in the last year (at least three sessions)
  3. Having at least one residual pocket ≥ 5 mm with and intra bony component at least ≥ 2 mm
  Exclusion criteria:
  1. Smoking more than ten cigarettes per day
  2. Pregnancy
  3. Irregular compliance during SPT in the last year; and systemic conditions or therapies known to affect the healing potential of periodontal tissues (e.g., uncontrolled diabetes, oncological conditions, immunosuppressant drugs).
  Interventions: Procedure: Cavitron ultrasonic surgical aspirator

INTERVENTIONS:
Procedure: Cavitron ultrasonic surgical aspirator — Cavitron Ultrasonic Surgical Aspirator (CUSA) has proven to be effective in biofilm disruption and cell stimulation . The hypothesis is that the employment of CUSA for non-surgical treatment of infrabony defects thanks to its abilities to disrupt, fragment and aspirate granulation tissue, will allow the formation of larger and more stable blood clot.
  According to the anatomy of the osseous sites, the sonotrode (Sonocare 300 by Söring GmbH, Justus-von-Liebig-Ring 2 -25451 Quickborn Germany) will be inserted both intrasulcularly and trans gingivally (smallest tip is 0,8 mm); intrasulcularly in the cases of three wall defects, and trans gingivally in cases of one to two wall defects .

SUMMARY:
The primary outcome of the present study will be assess the percentage of pocket closure and the secondary aim to evaluate the clinical performance in terms of clinical attachment level (CAL) gain, probing pocket depth (PPD) reduction and gingival recession (REC) after the use of cavitron ultrasonic surgical aspirator (CUSA) in deep infrabony defects.

Patients who were previously treated with active periodontal therapy followed by one year of supportive periodontal therapy (at least three sessions) will be additionally treated by the aid of CUSA. Subjects will be reviewed at 7 days, 15 days, 1 month, 3 months and 6 months. These sessions will include supra-gingival professional mechanical plaque removal (PMPR) through the use of erythritol powder plus 14 μm. Clinical measurements of the defects and X-ray with bite block will be taken at baseline and 3 and 6 months.

DETAILED DESCRIPTION:
This will be a Phase 2 non-controlled clinical trial performed on patients with infrabony defects to test whether the employment of CUSA for treating periodontal patients:

1. Provides benefits in terms of a PPD reduction and CAL gain
2. Is comfortable for patients and operators; and is free from adverse events

All subjects included in the study will be consecutive periodontal patients attending a private clinic in Settimo Milanese (Milan, Italy) who will be treated by two operators with similar experience in non surgical produce who performed a specific training for CUSA on a periodontal model.

The clinical procedure will be always performed in a single session. Before intervention, all cases will receive local anaesthesia with 1:100.000 mepivacaine.

All residual pockets ≥ 5 mm will be treated with

1. Ultrasonic debridement: to minimize trauma to the soft tissues, the investigators used piezo-electric devices with specific thin and delicate tips (E.M.S. Electro Medi- cal Systems S.A. Chemin de la Vuarpillière, 31 1260, Lyon Swizerland).
2. Flapless treatment: according to the anatomy of the osseous sites, the sonotrode (Sonocare 300 by Söring GmbH, Justus-von-Liebig-Ring 2 -25451 Quickborn Germany) will be inserted both intrasulcularly and trans gingivally (smallest tip is 0,8 mm); intrasulcularly in the cases of three wall defects, and trans gingivally in cases of one to two wall defects . The stack of piezo-electric quartzes transforms the electrical energy from the generator into a longitudinal, mechanical vibration of the sonotrode tip. When the tip of the sonotrode approaches the tissue, the ultrasonic energy, as a result of the high force of acceleration and cavitation effect, separates cells from the conglomerate of tissues (fragmentation). The fragmented tissue can be aspirated as a semiliquid substance through the sonotrode hole, freeing the defect from the formation of a stable blood clot.

   The end point will be achieving a condition in which the infrabony defect is free from the granulation tissue.
3. After CUSA treatment, to stimulate the formation of a stable blood clot, the use of any sub gingival rinses will be avoided.

No medications will be prescribed advising the patients to use painkillers (NSAIDs) if they experience postoperative pain.

Subjects will be reviewed at 7 days, 15 days, 1 month, 3 months and 6 months. These sessions will include supra-gingival professional mechanical plaque removal (PMPR) through the use of erythritol powder plus 14 μm (AIR-FLOW® MASTER -EMS).

Clinical measurements of the defects and X-ray with bite block will be taken at baseline and 3 and 6 months.

Outcomes :

* Pocket Closure proportion (PPD < 5 mm);
* Probing depth (PPD) reduction;
* CAL gain; and
* Gingival recession.
* Comfort and acceptability of the patient during and after the procedure, as measured by interviews, use of painkillers in the following three days and the visual analogue scale (VAS) after one week
* Comfort and convenience of the operator during the procedure, as measured by interviews at the end of the procedure; and adverse events

Continuous variables will be expressed as the mean ± standard deviation (SD). Dichotomous data will be expressed as a percentage. The comparison between baseline and 6 months after flapless treatment will be performed by applying a Wilcoxon signed ranked test.

ELIGIBILITY:
Inclusion Criteria:

1. Having received a diagnosis of chronic periodontitis (Armitage 1999)
2. Being treated by full mouth debridement, and supportive periodontal treatment (SPT) in the last year (at least three sessions) by one of the authors
3. Having at least one residual pocket ≥ 5 mm with and intra bony component at least ≥ 2 mm

Exclusion Criteria:

1. Smoking more than ten cigarettes per day
2. Pregnancy
3. Irregular compliance during SPT in the last year; and systemic conditions or therapies known to affect the healing potential of periodontal tissues (e.g., uncontrolled diabetes, oncological conditions, immunosuppressant drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Periodontal healing - Pocket Closure proportion | 6 months
  Periodontal Pocket Depth (PPD) is the measured distance from the free end of the gingival margin to the bottom of the periodontal pocket. PPD will be measured with the periodontal probe in millimeter (mm) and recorded in the periodontal charting. Successful result would be the achievement of residual PPD < 5 mm

SECONDARY OUTCOMES:
Comfort of the patient - Visual Analogue Scale (VAS) for pain | 1 week
  Comfort of the patient during and after the procedure will be measured by interviews, recording the 10 cm-long visual analogue scale (VAS) for pain, ranging from 0 to 10 cm, where is "no pain" 10 is "the worst pain perceivable".
Comfort of the patient by interview | 1 week
  Comfort of the patient during and after the procedure will be measured by interviews, using of painkillers in the following three days
Comfort of the operator | 1 day
  Comfort of the operator during the procedure will be recorded by interviews at the end of the procedure with a questionnaire
Adverse effects | 1 day
  Adverse effects of patients will be recorded via questionnaire
Clinical attachment level (CAL) gain | 6 months
  Clinical attachment level (CAL) is the distance from the cementoenamel junction to the bottom of the periodontal pocket. CAL gain will be measured with the periodontal probe in millimeter (mm), comparing CAL baseline to post-treatment values.
Gingival recession | 6 months
  Gingival recession is the displacement of the marginal tissue apical to the cemento-enamel junction, thus the distance from the cementoenamel junction to the free gingival margin. Gingival recession will be measured with the periodontal probe in millimeter (mm), comparing gingival recession baseline to post-treatment values.
Periodontal Pocket Depth (PPD) reduction | 6 months
  Periodontal Pocket Depth (PPD) reduction will be will be measured with the periodontal probe in millimeter (mm), comparing PPD baseline to post-treatment values.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Lodi, DMD, Principal Investigator — University of Milan
Locations (1):
- Studio Ghezzi, Settimo Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nibali L. Intrabony defects and non-surgical treatment. Prim Dent J. 2014 Aug;3(3):48-50. doi: 10.1308/205016814812736682. PMID 25198639
- [Background] Heitz-Mayfield LJ. How effective is surgical therapy compared with nonsurgical debridement? Periodontol 2000. 2005;37:72-87. doi: 10.1111/j.1600-0757.2004.03797.x. No abstract available. PMID 15655026
- [Background] El Moghazy WM, Hedaya MS, Kaido T, Egawa H, Uemoto S, Takada Y. Two different methods for donor hepatic transection: cavitron ultrasonic surgical aspirator with bipolar cautery versus cavitron ultrasonic surgical aspirator with radiofrequency coagulator-A randomized controlled trial. Liver Transpl. 2009 Jan;15(1):102-5. doi: 10.1002/lt.21658. PMID 19109835
- [Background] Brendan J. O'Dalya,b, Edmund Morrisb, Graham P. Gavinc, John M. O'Byrnea, Garrett B. McGuinnessb. High-power low-frequency ultrasound: A review of tissue dissection and ablation in medicine and surgery. Journal of Materials Processing Technology. Volume 200, Issues 1-3, Pages 38-58. 8 May 2008.
- [Derived] Ghezzi C, Donghi C, Ferrantino L, Varoni E, Lodi G. Ultrasonic Surgical Aspirator to Treat Deep Infrabony Defects: A New Flapless Minimally Invasive Approach. Adv Med. 2018 Jul 29;2018:3612359. doi: 10.1155/2018/3612359. eCollection 2018. PMID 30155496